CLINICAL TRIAL: NCT06412068
Title: A Prospective, Single-arm, Multi-center Exploratory Study on the First-line Treatment of Primary Mediastinal Large B-cell Lymphoma ( PMBCL ) With Sintilimab Combined With R-CHOP Regimen
Brief Title: A Prospective Study: Sintilimab and R-CHOP in PMBCL Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hua Wang, Associate senior doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-106
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Primary Mediastinal Large B Cell Lymphoma
Keywords: primary mediastinal large B cell lymphoma; sintilimab; R-CHOP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients diagnosed with PMBCL. (Experimental)
  Interventions: Drug: Combined anti-PD-1 and R-CHOP

INTERVENTIONS:
Drug: Combined anti-PD-1 and R-CHOP — Sintilimab,200mg, d1, intravenous drip; Rituximab,375mg／㎡, d1,intravenous drip; Cyclophosphamide,750mg／㎡,d2,intravenous drip; Doxorubicin,50mg／㎡ （or Liposome doxorubicin ，40 mg／㎡）,d2,intravenous drip; Vincristine,1.4mg／㎡, d2（Maximum dose 2mg),intravenous drip; Prednisone, 60mg/ m2 , d1-d5,oral administration.

SUMMARY:
The purpose of this multi-center, single arm, phase Ⅱ clinical trail is to evaluate the efficacy and toxicity of sintilimab combined with R-CHOP regimen as first-line treatment for primary mediastinal large B-cell Lymphoma (PMBCL)

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of PMBCL , and did not receive any previous treatment for PMBCL ;
* Predicted survival time ≥ 6 months ;
* 18-75 years ;
* IPI score 0-3；
* ECOG performance status 0-2 ;
* Clinicians judge that the patient is suitable for the treatment of primary mediastinal large B-cell lymphoma ;
* After the patient was enrolled in the trial, other drugs that may have therapeutic effects on primary mediastinal large B-cell lymphoma were not acceptable ;
* WBC ≥ 3 × 109 / L, NE ≥ 1.5 × 109 / L, PLT ≥ 100 × 109 / L ;
* Serum creatinine ≤ 1.5mg / dL, creatinine clearance rate ≥ 50mL / min ;
* ALT, AST ≤ 3 × ULN ( normal upper limit ) ; total bilirubin ≤ 2 × ULN ;
* Sign the informed consent.

Exclusion Criteria:

* Other malignant diseases except PMBCL were diagnosed within 5 years；·Participating in other interventional clinical studies, or has received chemotherapy, radiotherapy, immunotherapy or biotherapy for lymphoma；
* Known allergies to test drugs or any excipient component of these products；·Allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation has been performed；
* Women in pregnancy or lactation；
* Severe infectious diseases, such as HIV infection, untreated active hepatitis B, active hepatitis C；
* The researchers believe that there are other potential risks that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
complete remission (CR) | 2years
overall response rate (ORR) | 2 years
  The proportion of patients with a PR and CR

SECONDARY OUTCOMES:
overall survival (OS) | 2 years
  The time calculated from enrollment until death from any cause, with living patients censored at the last known survival date
progression survival (PFS) | 2 years
  The time from enrollment until tumor progression or death from any cause, whichever occurred first
bio-marker analysis | 2 years
  Correlation between programmed death-ligand 1 expression and efficacy